CLINICAL TRIAL: NCT04285151
Title: Evaluation of Nd:YAG Laser Hyaloidotomy for Management of Premacular Subhyaloid Hemorrhage in Eyes With Proliferative Diabetic Retinopathy
Brief Title: Nd:YAG Laser Hyaloidotomy for Premacular Hemorrhage in Diabetic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sharif Yousef El Emam, Clinical Associate Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUOR002
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Proliferative Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Nd:YAG laser Hyaloidotomy — Using the YAG laser for opening the posterior hyaloid in eyes with premacular hemorrhage, and evacuating the entrapped hemorrhage

SUMMARY:
Premacular Subhyaloid hemorrhage is a sudden profound loss of vision in eyes with proliferative diabetic retinopathy (PDR). Pars plana vitrectomy is the treatment of choice for premacular hemorrhage in eyes with proliferative changes. Nd:YAG laser hyaloidotomy has been used to evacuate the premacular hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Eyes with premacular subhyaloid hemorrhage of more than 3 disc diameters, involving the fovea.
* Eyes with proliferative diabetic retinopathy

Exclusion Criteria:

* Dense media opacity (corneal/cataract)
* Patients with bleeding tendency or on anti-coagulant drugs

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement | 1 week
  Testing VA after YAG laser

IPD SHARING:
Plan to Share IPD: No